CLINICAL TRIAL: NCT06202937
Title: The Effect of Mother-Baby Yoga on Fragile Baby Perception Syndrome, Maternal Attachment, Depression-Anxiety-Stress in Mothers
Brief Title: The Effect of Mother-Baby Yoga Baby Perception, Maternal Attachment,Depression-Anxiety-Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, EMİNE SARIKAMIŞ KALE, Phd student, Hasan Kalyoncu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2023/64
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Mother-Infant Interaction
Keywords: Mother-Baby Yoga; Fragile Baby Perception Syndrome; Maternal Attachment; Depression-Anxiety-Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mother baby yoga (Experimental): Mother-baby yoga will be held with the babies discharged from the neonatal intensive care unit and their mothers
  Interventions: Behavioral: Mother Baby Yoga
- control (Experimental): the control group received the usual care
  Interventions: Other: No intervention:control

INTERVENTIONS:
Behavioral: Mother Baby Yoga — Fragile Baby Perception Syndrome, Maternal Attachment, Depression-Anxiety-Stress Level
  Arms: mother baby yoga
Other: No intervention:control — the control group received the usual care
  Arms: control

SUMMARY:
The research will be carried out in a randomized controlled manner to determine the positive benefits of yoga for mothers and babies who have given birth preterm and have been discharged, and to determine its effect on Fragile Baby Perception Syndrome, maternal attachment, depression-anxiety-stress levels.

DETAILED DESCRIPTION:
The World Health Organization (WHO) defines preterm newborns as babies born alive before completing the 37th week of gestation, regardless of birth weight. While the preterm birth rate in the world is 10%, the preterm rate in live births in our country in 2021 has increased compared to previous years and has been determined as 12.2%. Preterm babies account for 35% of neonatal deaths worldwide. According to WHO, approximately 15 million babies are born preterm every year. Complications arising from preterm birth are the leading cause of mortality among children under 5 years of age. Again, according to WHO, 16% of neonatal (0-27 days) deaths are caused by preterm birth.Preterm babies face many problems at home after discharge. It is reported in the literature that preterm babies need special care after birth, that they may need to stay in the neonatal intensive care unit (NICU) for a long time, and that babies' stay in the hospital or NICU is traumatic for families . In a study comparing the parenting competencies of families with a preterm baby at home with the parenting competencies of families with a term baby, it was reported that parents with a preterm baby were less self-confident and preferred to watch as spectators rather than actively participating in the baby's care . In the study titled Permanent Postnatal Depression After Preterm Birth conducted by Kukreja et al., it was determined that postpartum psychological distress and stress continued in mothers who gave birth preterm in the 6th week after birth.As a result of the preterm baby being hospitalized in the NICU, the mother's separation from her baby and her inability to give him the care he desires increases anxiety and stress in the mother. The mother, who feels guilty for giving birth to her baby early, sees herself as inadequate and feels a lack of self-confidence and cannot pay enough attention to her baby. The stress experienced by mothers in the first days also negatively affects the mother-infant relationship and maternal attachment . Stressful situations that negatively affect attachment can also increase the risk of anxiety and depression in the mother. A mother's loving attachment to her baby is one of the most important elements that affects the healthy development of the child. If a secure attachment cannot be established between mother and baby, the risk of developing emotional, social, physical and mental problems in the baby increases. The healthier the mother's communication and interaction with her baby in the early period; The faster the feeling of motherhood will develop. Additionally, the mother's anxiety, stress and fear will decrease .

Another problem experienced in preterm babies is that the mother, who gave birth before completing the pregnancy process, may fear losing her baby at any time after being discharged from home . The mother may not touch her baby, thinking that it will harm her, or she may delay this process and make it difficult to participate in the baby's care. These situations cause mothers to have difficulties in their relationship with their preterm babies and in baby care, and Fragile Baby Syndrome, defined by mothers as sensitive babies, may develop.One of the practices that will support the mother and baby during this period is yoga practice. Yoga is the oldest system in the world that emphasizes the importance of body, mind and spiritual balance in human development. Yoga, although mostly seen as a physical pursuit, is also a physio-psychological and psycho-spiritual subject; It is a teaching that ensures the mental, emotional and spiritual maturation of individuals along with physical maturation. When yoga is practiced in a disciplined manner, it enables the individual to become aware of his soul by connecting with his body and mind. Yoga is a practice that not only reduces stress but can also direct one's emotions and thoughts. Instead of questioning the negative experiences of the person, they accept them as they are and help them cope. Yoga has a very important place in supporting mother-baby communication after birth. It has been seen in the literature review that yoga is generally good for a person's psychological health and has a positive effect on self-efficacy . It is known that this practice enables mothers to intuitively be in close contact with their bodies and emotions . In line with the studies conducted, mother-baby yoga practice; helps the woman adapt to the changes occurring in her body, during meditation.This is due to the fact that she communicates spiritually with her baby by touching her baby and making eye contact.It is thought that it may contribute to mother-infant bonding and change in the mother's perception of her baby, as a result of being able to cope with physiological and psychological stressors. It also has positive effects on the baby, such as increased growth and development, regular sleep, reduced stress, sensory, motor, mental and social development and many more.

The aim of the research was planned to consider the positive benefits of yoga for mothers and babies who had preterm birth and were discharged, and to examine its effect on depression, anxiety, stress level, mother-infant attachment levels and mothers' perception of fragility.

ELIGIBILITY:
Inclusion Criteria:

Baby;

* Born earlier than 37 weeks of gestation,
* Those who were treated in the neonatal intensive care unit and discharged at least 8 and at most 16 weeks ago,
* Does not have any chronic disease,
* No congenital defects,
* Babies who have been evaluated for Developmental Hip Dysplasia and have received approval from their physician to practice yoga.

Mother's;

* Speaks Turkish,
* Those who are over 18 years old,
* Having internet access at home
* No physical illness that prevents yoga
* Those who want to participate in the study voluntarily,
* Mothers who have been approved by their physician to do yoga

Exclusion Criteria:

* Their baby has a genetic disease or congenital disorder,

  * Mothers and babies who are declared unsuitable for yoga by the physician
  * Mothers who have not completed 10 courses or who wish to withdraw at any stage of the study

Ages: 2 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-02 (Actual)

PRIMARY OUTCOMES:
Fragile Infant Perception Scale | 8 weeks
  it is an assessment tool developed to evaulate Fragile Infant Perception The total score of the scale is 50. A score of 27 or above from the scale indicates that the perception of fragility is high.
Maternal Attachment Scale | 8 weeks
  The scale contains direct statements rated between 1-4 (never, sometimes, often, always). Scores between 26 and 104 are obtained from the scale. A higher score means higher maternal attachment.
Depression, Anxiety, Stress Scale (DASS-21 | 8 weeks
  0-3 point each item min 0 max 21 total point each subscale

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Emine Sarıkamış Kale, Batman, Merkez
  - Hasan Kalyoncu University, Gaziantep, Şahinbey

REFERENCES:
- [Derived] Koc Ozkan T, Cigdem Z, Sarikamis Kale E, Kale Y. The effect of mother-baby yoga on mother's depression-anxiety-stress levels, perception of fragile baby, and maternal bonding: A randomized controlled trial. J Pediatr Nurs. 2025 Nov-Dec;85:171-180. doi: 10.1016/j.pedn.2025.07.029. Epub 2025 Jul 31. PMID 40749378